CLINICAL TRIAL: NCT06115772
Title: Prospective Assessment of HPV Associated Anogenital Pathology in Female Patients and Female Partners of Patients With Confirmed HPV Associated Oropharyngeal Carcinoma (PAP-OP)
Brief Title: Prospective Assessment of HPV Associated Anogenital Pathology in Female Patients and Female Partners of Patients With Confirmed HPV Associated Oropharyngeal Carcinoma, PAP-OP Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-005420; NCI-2023-04392 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-005420 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Human Papillomavirus-Positive Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants complete surveys, watch an educational video on HPV vaccination and undergo collection of blood and saliva samples on study. Patients also undergo cervical screening per standard of care and may receive a referral to gynecology if not up to date on anogenital screening.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates how often women with throat (oropharyngeal) cancer or who have a partner with oropharyngeal cancer get anogenital infections with high risk, potentially cancer-causing types of human papilloma virus (HPV).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Prospectively determine the incidence of anogenital infection with high-risk HPV serotypes and HPV-associated anogenital lesions in female patients with newly diagnosed HPV(+)OPSCC and female partners of patients with HPV(+)OPSCC, and compare this with retrospective review of exams and paps obtained during routine well woman checks in Rochester MN.

II. To determine the risk of requiring additional procedures or treatments secondary to these diagnoses.

III. To determine the sexual health and well-being among patients and partners with HPV(+)OPSCC.

IV. To develop standardized patient education and recommendations for referral and screening for this patient population.

V. Measure patient satisfaction with study education and anogenital pathology screening process via internal questionnaire.

OUTLINE: This is an observational study.

Participants complete surveys, watch an educational video on HPV vaccination and undergo collection of blood and saliva samples on study. Patients also undergo cervical screening per standard of care and may receive a referral to gynecology if not up to date on anogenital screening.

ELIGIBILITY:
Inclusion Criteria:

* * Female patients with diagnosed HPV(+)OPSCC seen at the Mayo Clinic, Rochester

  * Age ≥ 18
  * Female partners of Mayo Clinic patients with diagnosed HPV(+)OPSCC
  * Patient has given permission to give his/her blood/saliva sample for research testing
  * Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* * HPV(-) OPSCC

  * Unable to provide informed consent
  * Unwilling to attend screening visit at Mayo Clinic site, if indicated
  * Unwilling/unable to complete surveys electronically

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients and female partners of patients with confirmed HPV associated oropharyngeal carcinoma (PAP-OP)
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and prevalence of HPV(+) associated anogenital pathology in patients with newly diagnosed HPV(+)OPSCC | Baseline (at enrollment)
  Prevalence and incidence of human papilloma virus (HPV)-related anogenital disease in female patients with HPV-mediated oropharyngeal squamous cell carcinoma (HPV(+)OPSCC) will be compared to a population of patients with similar demographic and comorbidity status. Rates will be compared across groups using tests for proportional variables (Fisher's exact, Chi Square).
Incidence and prevalence of HPV(+) associated anogenital pathology in partners of patients with newly diagnosed HPV(+)OPSCC | Baseline (at enrollment)
  Prevalence and incidence of human papilloma virus (HPV)-related anogenital disease in female partners of HPV-mediated oropharyngeal squamous cell carcinoma (HPV(+)OPSCC) patients will be compared to a population of patients with similar demographic and comorbidity status. Rates will be compared across groups using tests for proportional variables (Fisher's exact, Chi Square).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Van Abel, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials